CLINICAL TRIAL: NCT06808308
Title: Prognostic Value of PARS Classification in Predicting Post-recurrent Survival for Locally Recurrent Rectal Cancer Patients Undergoing Salvage Radical Surgery
Brief Title: Prognostic Value of PARS Classification for Locally Recurrent Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Zerong, Deputy Director of the Department, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2025ZSLYEC-050
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Local Recurrence of Malignant Tumor of Rectum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The pathological specimens before operation and the specimens after operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PARS Type I: Patients with central recurrence who had zero or one PHF were classified as PARS Type I.
- PARS Type II: Patients with central recurrence who had two and more PHFs were classified as PARS Type II. Central recurrences with two and more PHFs and non-central recurrences with no PHF were also classified as PARS Type II.
- PARS Type III: Patients with non-central recurrence who had one and more PHF were classified as PARS Type III

SUMMARY:
The aim of this retrospective study was to explore the predictors of post-recurrent survival in locally recurrent rectal cancer patients undergoing salvage radical surgery. Based on the identified risk factors, investigators propose a new risk stratification to facilitate the development of strategies for surgical treatment and follow-up care.

DETAILED DESCRIPTION:
With the introduction of total mesorectal excision (TME) and neoadjuvant chemoradiotherapy, the local recurrence rate of rectal cancer after surgery has markedly decreased; however, 5-18% of patients still experience recurrence in the pelvic field, significantly affecting their quality of life and contributing to high mortality rates. Several clinical and histologic features have been associated with the development of locally recurrent rectal cancer (LRRC), including higher primary T/N stage, positive margins, distal tumors, and histopathologic risk features such as tumor deposits (TD), lymphovascular invasion (LVI), and perineural invasion (PNI). Managing these recurrences is challenging, making risk stratification for re-recurrence through multidisciplinary evaluation essential for achieving personalized treatment in LRRC patients. Current imaging examinations typically stratify LRRC patients based on tumor recurrence patterns to guide clinical interventions. Due to primary treatment and varying local recurrence patterns, the pelvic fascial planes of LRRC patients are often altered or even absent, complicating surgery due to increased involvement of nearby organs or structures. Previous studies have indicated that surgical margin is the most crucial prognostic factor, with LRRC patients achieving R0 resections having a more favorable prognosis compared to those undergoing R1 or R2 resections or conservative treatments. Other potential features, such as gender, prior abdominoperineal resection, and advanced primary tumor stage, have been suggested to lead to poor post-recurrence prognoses; however, the prognostic impact of primary histologic risk features (TD, LVI, PNI) has rarely been addressed. Currently, there is no agreed-upon standardized treatment algorithm for LRRC, and nearly half of patients undergoing salvage radical surgery still experience re-recurrence within 12 months post-operation. The survival stratification of LRRC patients receiving salvage radical surgery remains underexplored.

ELIGIBILITY:
Inclusion Criteria:

* (1) the primary tumor was located in the sigmoid colon or rectum, following prior radical tumor resection;
* (2) local recurrence was confirmed through CT, MRI, and serum cancer biomarker test, or endoscopic biopsy;
* (3) the recurrent site was confined to the pelvis;
* (4) the recurrent tumor underwent R0 or R1 surgical resection;
* (5) the absence of uncontrollable distant metastases at the time of salvage radical surgery.

Exclusion Criteria:

* (1) patients with unresectable tumors identified before salvage radical surgery, leading to palliative therapy;
* (2) a recurrence interval of less than three months;
* (3) incomplete baseline characteristics, including pathologic data from the initial treatment;
* (4) loss to follow-up.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 865 LRRC patients were found in our hospital between January 2011 and December 2022. Finally, 199 patients diagnosed with LRRC who underwent salvage radical surgery were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
PRS | PRS was calculated from the date of salvage radical surgery until the date of death or until censored at the last follow-up, assessed up to 140 months.
  Post-recurrent survival

SECONDARY OUTCOMES:
DFS | DFS was calculated from the date of salvage radical surgery until the date when recurrence or metastasis was detected, assessed up to 140 months.
  Disease-free survival
LrRFS | LrRFS was calculated from the date of salvage radical surgery until the date when any local re-recurrence was detected by imaging or histology, or until censored at the last follow-up or death, assessed up to 140 months.
  Local re-recurrent free survival

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email